CLINICAL TRIAL: NCT02231944
Title: An Open Study to Investigate the Safety and Efficacy of Replenine®-VF in Severe Haemophilia B Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: R9VFSE
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

ARMS (1):
- Replenine®-VF (Experimental)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)

INTERVENTIONS:
Biological: Replenine®-VF (High Purity Factor IX)

SUMMARY:
To compare the first and second recovery assessments on Replenine®-VF and to evaluate recovery of different batches if patients changed batches during the study.

To evaluate Replenine®-VF in terms of long-term clinical efficacy, tolerance and safety

ELIGIBILITY:
Inclusion Criteria:

* Previously treated patients
* At least 12 years of age
* Severe Haemophilia B and without inhibitor to factor IX

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Recovery calculated from the first infusion of Replenine®-VF compared with that calculated 12 weeks later. | Baseline and 3 months post-baseline.
  Safety assessments included:
  * assessment of tolerance at injection site
  * assessment of Factor IX inhibitor development
  * assessment of frequency and type of adverse event
  * routine biochemistry and haematology at the start and end of Stage 1 and at the end of the study (Stage 2, if applicable)
  * screening for markers of viral infection at the start and end of each stage of the study (and if patients changed batches).

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (2):
  - Klinika Hematologii Instytutu Medycyny Wewnetrznej, Lodz
  - Klinika Hematologii AM Lublin, ul.Jaczewskiego 8, Lublin
- United Kingdom (5):
  - Addenbrooke's Hospital, Hills Road, Cambridge
  - University Hospital of Wales, Heath Park, Cardiff
  - The Royal London Hospital, London
  - Manchester Royal Infirmary, Oxford Road, Manchester
  - Norwich and Norfolk Hospital, Norwich

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk